CLINICAL TRIAL: NCT01832090
Title: Phase 4, Evaluation of Radiesse® Dermal Filler for Hand Treatment
Brief Title: Evaluation of Radiesse® Dermal Filler for Hand Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Merz Aesthetics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P110607
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Aging Hands
Keywords: aging; hands

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiesse® Injectable Dermal Filler (Experimental): Device: Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine-HCl)
  Interventions: Device: Radiesse® Injectable Dermal Filler
- Delayed Treatment (Active Comparator): Untreated controls crossed over to treatment with Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine) at 3 months
  Interventions: Device: Radiesse® Injectable Dermal Filler

INTERVENTIONS:
Device: Radiesse® Injectable Dermal Filler — Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Radiesse® Injectable Dermal Filler for hand treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, masked, controlled study to investigate the effectiveness of Radiesse® Dermal Filler for hand treatment, comprised of a 3-month main study followed by an open-label extension (OLEX) study through 12 months. At 3 months, untreated controls received Radiesse Dermal Filler for hand treatment and were followed for the remainder of the study. All study subjects were eligible for retreatment 6 months after initial treatment, and all subjects were followed through 12 months from study enrollment in the OLEX.

ELIGIBILITY:
Inclusion Criteria:

* Has right and left hands with rating of 2 or 3 on the Merz Hand Grading Scale (MHGS) as determined by a live, masked evaluator
* Is at least 18 years of age

Exclusion Criteria:

* Has history of hypertropic scarring
* Has a known bleeding disorder or receiving medication that will increase the risk of bleeding as the result of injection
* Has a known hypersensitivity to any of the components of Radiesse or local anesthesia
* Has received in past 6 months or plans to receive during the study dermal resurfacing procedure (chemical peel, dermabrasion, ablative laser resurfacing) or non-invasive skin tightening (Thermage®) in the dorsum of the hands
* Has received in past 2 weeks or plans to receive during the study prescription wrinkle therapies, topical steroids, skin irritating topical preparations, or pigmenting agents (self-tanning agents) in the dorsum of the hands
* Has had any dermal fillers or surgery in the dorsum of the hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Merz Investigative Site #004, San Diego, California
  - Merz Investigative Site #007, Vista, California
  - Merz Investigative Site #002, Garden City, New York
  - Merz Investigative Site #006, New York, New York
  - Merz Investigative Site #003, Nashville, Tennessee
  - Merz Investigative Site #001, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiesse® Injectable Dermal Filler: Device: Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine-HCl)
  Radiesse Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier
- Delayed Treatment: Untreated controls crossed over to treatment with Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine) at 3 months
  Radiesse Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier
Period: Overall Study
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Started | 89 | 29
Completed | 83 | 28
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Population: 113 of 114 subjects (99%) completed the main study through 3 months. One subject randomized to the control group suffered a non-study related broken hand after enrollment but prior to 3 month follow up and treatment. This subject's effectiveness data were imputed as "No change" for the purposes of the primary effectiveness analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment | Total
Number analyzed (Participants) | 85 | 29 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.0) | 54.8 (10.6) | 53.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 28 | 109
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 66 | 21 | 87
  African American | 3 | 3 | 6
  Hispanic | 12 | 3 | 15
  Asian | 3 | 1 | 4
  Other | 1 | 1 | 2
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick Skin Types (FST) represent a standard classification of skin color based on one's response to sun exposure (i.e., burns or tans), rather than defined by race or ethnicity.
  All FST were eligible for participation in the current study.
  See full FST descriptions in Astner S, Anderson RR. Skin phototypes 2003. J Invest Dermatol. 2004 Feb;122(2):xxx-xxxi.
  participants
    I: burns easily, never tans | 3 | 0 | 3
    II: burns easily, tans minimally with difficulty | 45 | 11 | 56
    III: burns moderately, tans moderately & uniformly | 19 | 11 | 30
    IV: burns minimally, tans moderately & easily | 13 | 4 | 17
    V: rarely burns, tans profusely | 4 | 2 | 6
    VI: never burns, tans profusely | 1 | 1 | 2
Hand Dominance [Number; unit: participants]
  Right | 79 | 26 | 105
  Left | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change on Merz Hand Grading Scale (MHGS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a mean change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by hand, among treated subjects and untreated controls. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: All primary effectiveness analyses were performed based on the intent-to-treat (ITT) population. This population includes all subjects randomized. One subject was randomized but did not receive treatment and was imputed as "No change" for the primary endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 85 | 29
Number analyzed (Hands) | 170 | 58
units on a scale
  Baseline | 2.6 (0.5) | 2.6 (0.5)
  3 Months | 1.5 (0.8) | 2.6 (0.5)
  Change from Baseline at 3 Months | -1.1 (0.9) | -0.1 (0.2)
Statistical Analysis 1: Comparison: Radiesse® Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: ≥ 1-point Change on the 5-point Merz Hand Grading Scale (MHGS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by hand, among treated subjects and untreated controls. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hands
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 85 | 29
Number analyzed (Hands) | 170 | 58
percentage of hands | 77.1 | 5.2
Statistical Analysis 1: Comparison: Radiesse® Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Primary Outcome: ≥ 1-point Change on the 5-point Merz Hand Grading Scale (MHGS), by Subject
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by subject, among treated subjects and untreated controls. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 85 | 29
percentage of participants | 75.3 | 3.4
Statistical Analysis 1: Comparison: Radiesse® Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Mean Change on Merz Hand Grading Scale (MHGS), by Hand, With Subjects Stratified by Age < 60 Years or ≥ 60 Years
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by mean change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by hand, among treated subjects and untreated controls, stratified by age < 60 years or ≥ 60 years. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: Single withdrawn subject imputed as "no change"
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Groups:
- Age < 60 and Radiesse® Injectable Dermal Filler; Age ≥ 60 and Radiesse® Injectable Dermal Filler: Device: Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine-HCl)
  Radiesse® Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.
- Age < 60 and Delayed Treatment; Age ≥ 60 and Delayed Treatment: Untreated controls crossed over to treatment with Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine) at 3 months
  Radiesse® Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.
Arm/Group | Age < 60 and Radiesse® Injectable Dermal Filler | Age < 60 and Delayed Treatment | Age ≥ 60 and Radiesse® Injectable Dermal Filler | Age ≥ 60 and Delayed Treatment
Number analyzed (Participants) | 67 | 18 | 18 | 11
Number analyzed (Hands) | 134 | 36 | 36 | 22
units on a scale
  Baseline | 2.5 (0.5) | 2.5 (0.5) | 2.7 (0.5) | 2.7 (0.5)
  3 Months | 1.4 (0.8) | 2.4 (0.5) | 1.7 (0.8) | 2.7 (0.5)
  Change from Baseline at 3 Months | -1.1 (0.9) | -0.1 (0.3) | -1.0 (0.8) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Age < 60 and Radiesse® Injectable Dermal Filler vs Age < 60 and Delayed Treatment vs Age ≥ 60 and Radiesse® Injectable Dermal Filler vs Age ≥ 60 and Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: ≥ 1-point Change on Merz Hand Grading Scale (MHGS), by Hand, With Subjects Stratified by Age < 60 Years or ≥ 60 Years
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by hand, among treated subjects and untreated controls, stratified by age < 60 years or ≥ 60 years. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: Single withdrawn subject imputed as "no change"
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hand
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 85 | 29
Number analyzed (Hand) | 170 | 58
percentage of hands
  Age < 60 years | 78.4 | 8.3
  Age ≥ 60 years | 72.2 | 0.0
Statistical Analysis 1: Comparison: Radiesse® Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p > 0.05, Fisher Exact

6. Secondary Outcome: ≥ 1-point Change on Merz Hand Grading Scale (MHGS), by Subject, With Subjects Stratified by Age < 60 Years or ≥ 60 Years
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3 months, by subject, among treated subjects and untreated controls, stratified by age < 60 years or ≥ 60 years. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: Single withdrawn subject imputed as "no change"
Measure: Number; unit: percentage of participants
Arm/Group | Radiesse® Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 85 | 29
percentage of participants
  Age < 60 years | 76.1 | 5.6
  Age ≥ 60 years | 72.2 | 0.0
Statistical Analysis 1: Comparison: Radiesse® Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p > 0.05, Fisher Exact

7. Secondary Outcome: Evenness in the Left Hand Versus the Right Hand Using the Merz Hand Grading Scale (MHGS) Among the Original Treatment Group Only
Description: To evaluate the efficacy of Radiesse for hand treatment by comparing the evenness in the left hand versus the right hand at 3 months using the 5-point Merz Hand Grading Scale (MHGS) among the original treatment group only. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3 months from baseline
Population: Single withdrawn subject imputed as "no change"
Measure: Number; unit: percentage of participants
Arm/Group | Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 85
percentage of participants
  0 points | 84.7
  1 point | 15.3
  > 1 point | 0

8. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings Among the Original Treatment Group Only
Description: To evaluate the efficacy of Radiesse for hand treatment by evaluating subject-reported, live Global Aesthetic Improvement Scale (GAIS) ratings at 3 months when compared to baseline among the original treatment group only
Time Frame: 3 months from baseline
Population: Single withdrawn subject imputed as "no change"
Measure: Number; unit: percentage of participants
Units Other Than Participants: Hands
Arm/Group | Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 85
Number analyzed (Hands) | 170
percentage of participants
  Very Much Improved | 31.8
  Much Improved | 44.1
  Improved | 21.8
  No Change | 2.4
  Worse | 0.0
  Total: At least "Improved" | 97.6

9. Secondary Outcome: Mean Change on the Merz Hand Grading Scale (MHGS), by Hand, Among All Treated Subjects Without Retreatment
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by mean change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3, 6, 9, and 12 months, by hand, among all treated subjects without retreatment. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Single withdrawn subject did not receive treatment and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Groups:
- Baseline: Radiesse® Injectable Dermal Filler; 3 Months Post-treatment: Radiesse® Injectable Dermal Filler; 6 Months Post-treatment: Radiesse® Injectable Dermal Filler; 9 Months Post-treatment: Radiesse® Injectable Dermal Filler; 12 Months Post-treatment: Radiesse® Injectable Dermal Filler: Device: Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine-HCl)
  Radiesse® Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.
Arm/Group | Baseline: Radiesse® Injectable Dermal Filler | 3 Months Post-treatment: Radiesse® Injectable Dermal Filler | 6 Months Post-treatment: Radiesse® Injectable Dermal Filler | 9 Months Post-treatment: Radiesse® Injectable Dermal Filler | 12 Months Post-treatment: Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 36 | 36 | 36 | 36 | 23
Number analyzed (Hands) | 72 | 72 | 72 | 72 | 46
units on a scale | 2.5 (0.5) | 1.3 (0.8) | 1.3 (0.9) | 1.4 (0.8) | 1.7 (0.8)
Statistical Analysis 1: Comparison: Baseline: Radiesse® Injectable Dermal Filler vs 3 Months Post-treatment: Radiesse® Injectable Dermal Filler vs 6 Months Post-treatment: Radiesse® Injectable Dermal Filler vs 9 Months Post-treatment: Radiesse® Injectable Dermal Filler vs 12 Months Post-treatment: Radiesse® Injectable Dermal Filler; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Mean Change on the Merz Hand Grading Scale (MHGS), by Hand, Among All Treated Subjects With Retreatment
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by mean change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3, 6, 9, and 12 months, by hand, among all treated subjects receiving retreatment. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Single withdrawn subject did not receive treatment and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Groups:
- 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler; 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler: Device: Radiesse Dermal Filler mixed with 2% lidocaine-HCl (final concentration: 0.3% lidocaine-HCl)
  Radiesse® Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.
Arm/Group | Baseline: Radiesse® Injectable Dermal Filler | 3 Months Post-treatment: Radiesse® Injectable Dermal Filler | 6 Months Post-treatment: Radiesse® Injectable Dermal Filler | 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 77 | 77 | 77 | 77 | 60
Number analyzed (Hands) | 154 | 154 | 154 | 154 | 120
units on a scale | 2.6 (0.5) | 1.5 (0.8) | 1.7 (0.7) | 1.4 (0.7) | 1.3 (0.6)
Statistical Analysis 1: Comparison: Baseline: Radiesse® Injectable Dermal Filler vs 3 Months Post-treatment: Radiesse® Injectable Dermal Filler vs 6 Months Post-treatment: Radiesse® Injectable Dermal Filler vs 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler vs 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: ≥ 1-point Change on the Merz Hand Grading Scale (MHGS), by Hand, Among All Treated Subjects With and Without Retreatment
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3, 6, 9 and 12 months, by hand, among treated subjects with and without retreatment. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Single withdrawn subject did not receive treatment and is not included in this analysis.
Measure: Number; unit: % hands with ≥ 1 point MHGS change
Units Other Than Participants: Hands
Arm/Group | 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 9 Months Post-treatment: Radiesse® Injectable Dermal Filler | 12 Months Post-treatment: Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 77 | 60 | 36 | 23
Number analyzed (Hands) | 154 | 120 | 72 | 46
% hands with ≥ 1 point MHGS change | 83.1 | 88.3 | 73.6 | 71.7

12. Secondary Outcome: ≥ 1-point Change on the Merz Hand Grading Scale (MHGS), by Subject, Among All Treated Subjects With and Without Retreatment
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by ≥ 1-point change on the 5-point Merz Hand Grading Scale (MHGS) between baseline and 3, 6, 9, and 12 months, by subject, among treated subjects with and without retreatment. A measure of successful or improved treatment effect is demonstrated by a decrease in MHGS score.
  MHGS categories are as follows:
  0 = no loss of fatty tissue;
  1 = mild loss of fatty tissue; slight visibility of veins; 3 = moderate loss of fatty tissue; mild visibility of veins and tendons; 4 = severe loss of fatty tissue; moderate visibility of veins and tendons; and 5 = very severe loss of fatty tissue; marked visibility of veins and tendons.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Single withdrawn subject did not receive treatment and is not included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 9 Months Post-treatment: Radiesse® Injectable Dermal Filler | 12 Months Post-treatment: Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 78 | 61 | 35 | 22
percentage of participants | 82.1 | 88.5 | 71.4 | 68.2

13. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings, by Subject, Among All Treated Subjects With and Without Retreatment
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by live, subject-completed Global Aesthetic Improvement Scale (GAIS) scores between baseline and 3, 6, 9, and 12 months, by subject, among treated subjects with and without retreatment
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Single withdrawn subject did not receive treatment and is not included in this analysis.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Hands
Arm/Group | 3 Months Post-treatment: Radiesse® Injectable Dermal Filler | 6 Months Post-treatment: Radiesse® Injectable Dermal Filler | 9 Months Post-treatment: Radiesse® Injectable Dermal Filler | 12 Months Post-treatment: Radiesse® Injectable Dermal Filler | 3 Months Post-retreatment: Radiesse® Injectable Dermal Filler | 6 Months Post-retreatment: Radiesse® Injectable Dermal Filler
Number analyzed (Participants) | 113 | 113 | 35 | 22 | 77 | 61
Number analyzed (Hands) | 226 | 226 | 70 | 44 | 154 | 122
percentage of participants
  Very Much Improved | 29.2 | 41.6 | 32.9 | 11.4 | 44.2 | 43.4
  Much Improved | 44.7 | 30.5 | 34.3 | 40.9 | 39.0 | 24.6
  Improved | 24.3 | 21.2 | 27.1 | 34.1 | 15.6 | 27.0
  No Change | 1.8 | 6.6 | 5.7 | 13.6 | 1.3 | 4.9
  Worse | 0 | 0 | 0 | 0 | 0 | 0
  Total: At least "Improved" | 98.2 | 93.4 | 94.3 | 86.4 | 98.7 | 95.1

ADVERSE EVENTS:
Description: 113 of 114 subjects (99%) completed the main study through 3 months. One subject randomized to the control group suffered a non-study related broken hand after enrollment but prior to 3 month follow up and treatment. This subject's effectiveness data were imputed as "No change" for the purposes of the primary effectiveness analysis.
Arm/Group | Radiesse® Injectable Dermal Filler
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 50/113
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiesse® Injectable Dermal Filler (N=113)
Bruising (Skin and subcutaneous tissue disorders) | 21
Swelling (Skin and subcutaneous tissue disorders) | 23
Redness (Skin and subcutaneous tissue disorders) | 9
Itching (Skin and subcutaneous tissue disorders) | 4
Pain (Skin and subcutaneous tissue disorders) | 7
Nodule, Bumps/Lumps (Skin and subcutaneous tissue disorders) | 7
Other, not within pre-defined (expected) AE categories (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No